CLINICAL TRIAL: NCT00734942
Title: Improved Health-Related Quality of Life for Young Carers and Their Families in Germany on the Basis of Evidence-Based Family-Oriented Support
Brief Title: Development and Implementation of Evidence-Based Family-Oriented Support for Young Carers and Their Families in Germany
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Witten/Herdecke (Other)
Responsible Party: Prof. Dr. Wilfried Schnepp, Universität Witten/Herdecke
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 01GT0619
Record Dates: First submitted 2008-08-12; First posted 2008-08-14 (Estimated); Last update posted 2008-12-23 (Estimated); Status verified 2008-08

CONDITIONS: Chronic Illness
Keywords: young carers; family support; children (up to the age of 18) of chronically ill parents
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): intervention group
  Interventions: Other: support service
- 2 (No Intervention): waiting group

INTERVENTIONS:
Other: support service — * professional partners for communication
  * befriending with other families concerned
  * information and education (about illness, symptoms, first aid, caring)
  * free-time activities and time out
  * homework assistance
  * administrative advise
  * support for everyday life
  Arms: 1

SUMMARY:
The purpose of this study is to develop and implement evidence-based and family-oriented support for young carers and their families in Germany. Hypothesis is that families' own support mechanisms, combined with externally provided support that is determined by the families' specific needs, will help to overcome their burden and enable families to live in the way they wish to despite chronic illness. This will lead to a measurable increase in HRQOL of children concerned.

ELIGIBILITY:
Inclusion Criteria:

* children of mentally ill parents (chronic illness)
* children of somatically ill parents (chronic illness)

Exclusion Criteria:

* children of drug addicted parents

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 150 (Estimated)
Dates: Start 2009-01; Primary Completion 2009-12 (Estimated); Study Completion 2010-03 (Estimated)

PRIMARY OUTCOMES:
health-related Quality of Life in children | study start and after 5 month of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Metzing-Blau, Dr., Principal Investigator — Institute of Nursing Science; Witten/Herdecke University; Wilfried Schnepp, Prof.Dr., Study Director — Institute of Nursing Science; Witten/Herdecke University
Locations (1):
- Institute of Nursing Science, Witten, North Rhine-Westphalia, Germany

REFERENCES:
- [Background] Metzing S, Schnepp W. [The impact of caring on young carer's lives. An international literature review (1990-2006)]. Pflege. 2007 Dec;20(6):331-6. doi: 10.1024/1012-5302.20.6.331. German. PMID 18357746
- [Background] Sabine M, Schnepp W. [Children and adolescents as caregivers: who they are and what they do. An international literature review (1990-2006)]. Pflege. 2007 Dec;20(6):323-30. doi: 10.1024/1012-5302.20.6.323. German. PMID 18357745
- [Background] Schlarmann JG, Metzing-Blau S, Schnepp W. The use of health-related quality of life (HRQOL) in children and adolescents as an outcome criterion to evaluate family oriented support for young carers in Germany: an integrative review of the literature. BMC Public Health. 2008 Dec 17;8:414. doi: 10.1186/1471-2458-8-414. PMID 19091099
- [Derived] Schlarmann JG, Metzing S, Schoppmann S, Schnepp W. Germany's First Young Carers Project's Impact on the Children: Relieving the Entire Family. A Qualitative Evaluation. Open Nurs J. 2011;5:86-94. doi: 10.2174/1874434601105010086. Epub 2011 Oct 26. PMID 22135716
- See also: Website of the study — http://www.kinder-kranker-eltern.de